CLINICAL TRIAL: NCT05942664
Title: Can Habitual Sleeping Habits Predict Performance Outcomes Following Sleep Deprivation?
Brief Title: Sleeping Habits on Performance Following Sleep Deprivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Philip Millar, Associate Professor, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 23-01-019
Record Dates: First submitted 2023-06-26; First posted 2023-07-12 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Sleep; Athletic Performance; Hemodynamics
Keywords: Sleep habits; Chronotype; Sleep quality; Cycling time trial performance
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Sleep

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants and investigators are blinded to power output during the time trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal sleep (Sham Comparator): Participants will be asked to sleep during their normal sleep times prior to this visit
  Interventions: Behavioral: Sleep
- Sleep deprivation (Active Comparator): Participants will be asked to go to bed normally but wake up earlier, such that normal sleep duration is restricted by 60%. For example, if someone normally sleeps for 8 hours by falling asleep at 11 pm and waking up at 7 am, they will be asked to fall asleep normally (11 pm) and sleep for 3.2 hours, which results in a wake-up time of 2:12 am.
  Interventions: Behavioral: Sleep

INTERVENTIONS:
Behavioral: Sleep — Sleep will be restricted to 60% normal sleep duration

SUMMARY:
The goal of this randomized crossover clinical trial is to determine if habitual sleeping habits can predict endurance performance following a night of partial sleep deprivation in healthy untrained, recreationally trained, and trained cyclists (18-50 years, ~50% females). The main questions it aims to answer are:

1. Can habitual sleeping habits predict, or do different types of sleepers alter, performance outcomes following sleep deprivation?
2. Does sleep deprivation alter blood pressure, heart rate, or metabolic responses during a 20-minute time trial, and/or are these altered amongst different types of sleepers?

   * Participants will be asked to perform 4 performance tests (20-minute time trial), 2 for familiarization, and 2 testing visits (1 under normal sleep and 1 under partial sleep deprivation).
   * For 1 week prior to each testing visit, sleep will be tracked using an ActiGraph device.

The investigators hypothesize that habitual early sleepers, poor sleepers, those with greater variability in sleep duration, and females will show the greatest impairments in performance following partial sleep deprivation.

DETAILED DESCRIPTION:
Five separate visits will take place. Participants will be asked to abstain from heavy exercise, napping, alcohol, recreational drugs, and acute supplementation or medication use (i.e., melatonin, antihistamines) 24 hours before each visit. The first visit will always be the introductory visit, which will be followed by two familiarization visits. The next two visits will be testing visits and randomized (one normal sleep visit and one sleep deprivation visit).

Introductory visit: Prior to arriving at the lab, participants will read over and sign the consent form, complete the Pittsburgh Sleep Quality Index (PSQI), complete the Morningness-Eveningness Questionnaire (MEQ), complete a general health questionnaire, and complete the PAR-Q+ remotely. After obtaining consent and upon arriving at the lab, height and weight will be measured. This will be followed by a maximal exercise test to assess peak oxygen uptake (VO2peak) on a cycle ergometer. After this, participants will be given a rest period, which will be followed by the completion of a 5-minute time trial so the participant can get familiarized with pushing themselves during the performance test.

Pre-testing: Participants will be equipped with an ActiGraph device to measure sleeping patterns over a 1-week time frame prior to each testing visit as well as the night prior to each familiarization visit. These data will then be used to determine each participant's sleep-wake schedule for the testing visits. Furthermore, the day prior to each familiarization visit and testing visit, participants will be asked to complete a food diary using an online app (MyFitnessPal), which will ask participants to list the ingredients and quantity of each ingredient consumed for each meal and beverage that day, night and subsequent day. Participants will be asked to abstain from food for 4 hours upon arriving at the lab, prior to each familiarization and testing visit.

Familiarization visits: Upon lab arrival, participants will be provided with a standardized snack, which includes instant Quaker oats mixed with water. The amount will be based on body weight (1 gram of carbohydrates per body weight in kilograms). Following this, the participant will complete a 20-minute time trial on a cycle ergometer.

Testing visits: Upon lab arrival, participants will lay supine quietly, and resting hemodynamic measurements (blood pressure and heart rate) will commence. Following this, participants will consume the same standardized snack as the familiarization visit, and then a 20-minute time trial on a cycle ergometer.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-50 years
* Free of known cardiovascular or metabolic diseases or sleep disorders
* No history of smoking (within the past 3 months)
* Able to engage in physical activity assessed through the physical activity readiness questionnaire (PAR-Q+) (answer no to all questions
* No prescription of chronic medications other than oral contraceptives
* Able to abide by sleep protocols for all visits
* Individuals who are able to consume the ingredients of instant oatmeal (whole grain oats, sugar, salt, and natural flavour)
* Individuals who are not pregnant

Exclusion Criteria:

* Ages <18 years, >50
* Individuals diagnosed with cardiovascular or metabolic disease or sleep disorders
* Has a history of smoking (within the past 3 months)
* Not ready to engage in physical activity (answer yes to one or more questions in PAR-Q+)
* Individuals with prescription of chronic medications other than oral contraceptives
* Unable to abide by sleep protocols for any testing visit
* Individuals who are unable to consume the ingredients of instant oatmeal (whole grain oats, sugar, salt, and natural flavour)
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Performance | During each familiarization visit and testing visit (4 time points total)
  Mean power achieved during a 20-minute time trial on a cycle ergometer

OTHER OUTCOMES:
Resting systolic and diastolic blood pressure | During both testing visits (2 time points total)
  Resting blood pressure while participant is supine, assessed in 1-minute intervals through an automated oscillometric device and non-invasive, continuous blood pressure (i.e., on a heartbeat-by-beat basis)
Resting heart rate | During both testing visits (2 time points total)
  resting heart rate while participant is supine, assessed via ECG
Systolic and diastolic blood pressure during exercise | During the introductory visit and during each familiarization visit and testing visit (5 time points total)
  Blood pressure during the VO2peak test, 12-minute warm up, and performance tests, in 2-minute intervals, assessed using an automated oscillometric device
Heart rate during exercise | During the introductory visit and during each familiarization visit and testing visit (5 time points total)
  Heart rate during the VO2peak test, 12-minute warm up, and performance tests, on a heartbeat-by-beat basis, assessed using a heart rate monitor
Gross efficiency during exercise | During each familiarization visit and testing visit (4 time points total)
  Movement efficiency during the 12-minute warm up, prior to the performance tests. This will be calculated using the following formula: (work (J)/energy expenditure (J))*100. Work is calculated as: (watts during the warm up * time) and energy production is determined by the metabolic cart, and will be further broken down into joules by multiplying energy expenditure in kcals by 4184.
Oxygen uptake during exercise | During the introductory visit and during each familiarization visit and testing visit (5 time points total)
  Oxygen uptake during the VO2peak test, 12-minute warm up, and performance tests, assessed on a breath-by-breath basis using a metabolic cart
Carbon dioxide production during exercise | During the introductory visit and during each familiarization visit and testing visit (5 time points total)
  Carbon dioxide production during the VO2peak test, 12-minute warm up, and performance tests, assessed on a breath-by-breath basis using a metabolic cart
Systolic and diastolic blood pressure during recovery | During each familiarization visit and testing visit (4 time points total)
  Three minutes of recovery blood pressure following the performance tests, in 1-minute intervals
Heart rate during recovery | During each familiarization visit and testing visit (4 time points total)
  Three minutes of heart rate following the performance tests, on a heartbeat-by-beat basis, assessed using a heart rate monitor
Oxygen uptake during recovery | During each familiarization visit and testing visit (4 time points total)
  Three minutes of oxygen uptake following the performance tests, assessed breath-by-breath, using a metabolic cart
Carbon dioxide production during recovery | During each familiarization visit and testing visit (4 time points total)
  Three minutes of carbon dioxide production following the performance tests, assessed breath-by-breath, using a metabolic cart

CONTACTS AND LOCATIONS:
Overall Officials: Philip Millar, Principal Investigator — University of Guelph
Locations (1):
- University of Guelph - Human Cardiovascular Physiology Laboratory, Guelph, Ontario, Canada